CLINICAL TRIAL: NCT03333213
Title: Gua Sha Therapy for Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Gua Sha Therapy for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research Director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-3594
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gua Sha therapy (Experimental): Patients' backs were first covered with Tumarol N Balsam. The study physician then applied a round-edged instrument (the inside smooth edged lip of a metal cap) to patients' skin in downward strokes. Patients were treated twice with a 7-day interval.
  Interventions: Other: Gua Sha
- Waitlist control group (No Intervention): Treatments in the control group were not regulated but patients were asked to continue their self-directed medical care. They were offered the Gua Sha therapy once the trial was concluded.

INTERVENTIONS:
Other: Gua Sha
  Arms: Gua Sha therapy

SUMMARY:
Chronic low back pain is a major public health burden with only limited evidence of effectiveness for complementary and traditional therapies. Gua Sha is a traditional East Asian therapy traditionally used in the treatment of spinal pain. This study aimed to test the efficacy of Gua Sha therapy in patients with chronic low back pain A total of 50 patients with chronic low back pain were randomized to either two Gua Sha treatments (n=25) or a waitlist control group (n=25). Primary outcome measure was current pain intensity on a 100-mm visual analog scale; secondary outcome measures included back-related function (Oswestry Disability Index), movement-related pain (modified Pain on Movement Questionnaire), as well as pressure pain threshold, mechanical detection threshold, and vibration detection threshold.

DETAILED DESCRIPTION:
Chronic low back pain is a major public health burden with only limited evidence of effectiveness for complementary and traditional therapies. Gua Sha is a traditional East Asian therapy traditionally used in the treatment of spinal pain. This study aimed to test the efficacy of Gua Sha therapy in patients with chronic low back pain A total of 50 patients with chronic low back pain were randomized to either two Gua Sha treatments (n=25) or a waitlist control group (n=25). Primary outcome measure was current pain intensity on a 100-mm visual analog scale; secondary outcome measures included back-related function (Oswestry Disability Index), movement-related pain (modified Pain on Movement Questionnaire), as well as pressure pain threshold, mechanical detection threshold, and vibration detection threshold.

ELIGIBILITY:
Inclusion Criteria:

* non-specific low back pain at least once weekly for at least the previous 3 months
* average back pain intensity hat least 40mm on a 100mm visual analog scale (VAS)

Exclusion Criteria:

* specific low back pain due to trauma, disc protrusion, whiplash, congenital deformity of the spine, spinal stenosis, neoplasm, inflammatory rheumatic disease, or oncologic disease
* dystonia
* pregnancy
* invasive treatment of the spine or spinal surgery within the previous 4 weeks
* oral steroids or anticoagulants
* hemophilia or a skin condition in the area to be treated
* started a new treatment for low back pain within the previous month or planning to start a new treatment within the next month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 12 weeks
  100-mm visual analogue scale (VAS) ranging from 0mm meaning 'no pain at all' to 100mm meaning 'the worst pain imaginable'

SECONDARY OUTCOMES:
Pain on movement | 12 weeks
  Pain on Movement Questionnaire (POM)
Functional disability | 12 weeks
  Oswestry Disability Index (ODI)
Pressure-pain threshold (PPT) | 12 weeks
  PPT was measured using a digital algometer (Somedic AB, Horby, Sweden).
Mechanical detection threshold (MDT) | 12 weeks
  MDT was measured with a set of von Frey filaments (Somedic Sales AB, Horby, Sweden).
Vibration detection threshold (VDT) | 12 weeks
  VDT was determined using a Rydel-Seiffer tuning fork (64 Hz, 8/8 scale)
Adverse events | 12 weeks

IPD SHARING:
Plan to Share IPD: No